CLINICAL TRIAL: NCT01323777
Title: Clinical Investigation of AcrySof® IQ ReSTOR® Multifocal Toric Intraocular Lens Models SND1T3/ SND1T4/ SND1T5/ SND1T6
Brief Title: AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric Intraocular Lens (IOL) Clinical Study in Japan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J-10-050
Record Dates: First submitted 2011-03-24; First posted 2011-03-28 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-03

CONDITIONS: Cataracts
Keywords: Cataracts; Intraocular lens; Multifocal; Toric; Astigmatism; Presbyopia
MeSH Terms: conditions — Cataract; Astigmatism; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ReSTOR +3.0 (Experimental): AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL, model determined by preoperative keratometric astigmatism, bilateral implantation
  Interventions: Device: AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL

INTERVENTIONS:
Device: AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL — Multifocal IOL with extended secondary focal point and astigmatism correction implanted for long-term use over the lifetime of the cataract patient
  Other Names: Models SND1T3, SND1T4, SND1T5, SND1T6

SUMMARY:
The purpose of this study is to evaluate safety and effectiveness of AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL Models SND1T3, SND1T4, SND1T5, and SND1T6 when implanted to replace the natural lens in Japanese cataract patients.

DETAILED DESCRIPTION:
Eligible participants completed a preoperative examination of both eyes, implantation of the IOL at the operative visit for each eye, and up to 8 postoperative visits: Day 1-2, Day 7-14, and Day 30-60 after each implantation, and Day 120-180 and Day 330-420 after second eye implantation. The second implantation occurred within 30 days of the first.The primary eye was defined as the eye with higher astigmatism, with the other eye defined as the secondary eye. If both eyes had the same level of astigmatism, the first implanted eye was set as the primary eye.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent;
* Diagnosed with bilateral cataracts;
* Planned cataract removal by phacoemulsification;
* Potential postoperative visual acuity of 0.6 decimal or better in both eyes;
* Preoperative astigmatism ≥ 0.75 diopter;
* Clear intraocular media other than cataract in study eyes;
* Calculated lens power and astigmatism within the available range;
* Pupil size greater than or equal to 6 mm after dilation;
* Able to undergo second eye surgery within 30 days of the first eye surgery;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Irregular corneal aberration as demonstrated by corneal topography;
* Any inflammation or edema (swelling) of the cornea;
* Diagnosed degenerative visual disorders predicted to cause future acuity losses to a level worse than 0.6 decimal;
* Diabetic retinopathy;
* Previous refractive surgery, retinal detachment, corneal transplant;
* Glaucoma;
* Pregnant, nursing, or suspected of being pregnant;
* Currently participating in another investigational drug or device study;
* Other protocol-defined exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Group Manager, Surgical, Study Director — Alcon Japan, Ltd.
Locations (2):
- Japan (2):
  - Tokyo Dental College Suidobashi Hospital, Chiyoda-ku, Tokyo
  - Hayashi Eye Hospital, Fukuoka

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 2 study sites located in Japan.
Pre-assignment Details: This reporting group includes all implanted subjects (65).
Period: Overall Study
Arm/Group | ReSTOR +3.0
Started | 65
Completed | 65
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all implanted subjects.
Arm/Group | ReSTOR +3.0
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (9.9)
Age, Customized [Number; unit: participants]
  <60 years | 12
  60-69 years | 24
  70-79 years | 25
  ≥ 80 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 15
Region of Enrollment [Number; unit: participants]
  Japan | 65

OUTCOME MEASURES:

1. Primary Outcome: Monocular Uncorrected Distance Decimal Visual Acuity
Description: Visual acuity (VA) was tested monocularly (each eye separately) unaided at a distance of 5 meters (m) using a chart. VA was measured in decimal, with 1.0 decimal corresponding to 20/20 Snellen. A higher numeric value represents better visual acuity.
Time Frame: Day 1-2, Day 7-14, Day 30-60, Day 120-180, Day 330-420
Population: This analysis population includes all implanted subjects.
Measure: Number; unit: participants
Groups:
- Day 1-2; Day 7-14; Day 30-60; Day 120-180; Day 330-420: AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL, model determined by preoperative keratometric astigmatism
Arm/Group | Day 1-2 | Day 7-14 | Day 30-60 | Day 120-180 | Day 330-420
Number analyzed (Participants) | 65 | 65 | 65 | 65 | 65
participants
  Primary eye worse than 0.5 decimal | 3 | 3 | 1 | 0 | 1
  Primary eye 0.5 to less than 0.7 decimal | 12 | 4 | 6 | 3 | 5
  Primary eye 0.7 to less than 1.0 decimal | 29 | 27 | 30 | 27 | 28
  Primary eye 1.0 decimal or better | 21 | 31 | 28 | 35 | 31
  Secondary eye worse than 0.5 decimal | 5 | 1 | 3 | 1 | 0
  Secondary eye 0.5 to less than 0.7 decimal | 14 | 7 | 2 | 6 | 6
  Secondary eye 0.7 to less than 1.0 decimal | 21 | 22 | 28 | 28 | 27
  Secondary eye 1.0 decimal or better | 25 | 35 | 32 | 30 | 32

2. Primary Outcome: Monocular Uncorrected Near Decimal VA
Description: VA was tested monocularly unaided at a distance of 40 centimeters (cm) using a chart. VA was measured in decimal, with 1.0 decimal corresponding to 20/20 Snellen. A higher numeric value represents better visual acuity.
Time Frame: Day 30-60, Day 120-180, Day 330-420
Population: This analysis population includes all implanted subjects.
Measure: Number; unit: participants
Arm/Group | Day 30-60 | Day 120-180 | Day 330-420
Number analyzed (Participants) | 65 | 65 | 65
participants
  Primary eye worse than 0.4 decimal | 1 | 0 | 1
  Primary eye 0.4 decimal or better | 64 | 65 | 64
  Secondary eye worse than 0.4 decimal | 1 | 1 | 0
  Secondary eye 0.4 decimal or better | 64 | 64 | 65

ADVERSE EVENTS:
Time Frame: This reporting group includes all implanted subjects.
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a subject, user or other persons regardless of whether or not the event has a causal relationship with the medical device(s) or test procedure(s) in the study. AEs were collected as solicited comments from the subject and as observations by the study Investigator as outlined in the protocol.
Arm/Group | ReSTOR +3.0
Serious Adverse Events (participants affected / at risk) | 8/65
Other Adverse Events (participants affected / at risk) | 0/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ReSTOR +3.0 (N=65)
Atrial fibrillation paroxysmal (Cardiac disorders) | 1
Endophthalmitis (Primary Eye) (Infections and infestations) | 1
Eighth rib fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Gonarthrosis (Musculoskeletal and connective tissue disorders) | 1
Carcinoma hepatocellular (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Secondary surgical intervention (Primary Eye) (Surgical and medical procedures) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.